CLINICAL TRIAL: NCT05274256
Title: Implant Placement in Horizontally Deficient Maxillary Aesthetic Zone With Simultaneous Soft Tissue Augmentation Using De-epithelialized Free Gingival Graft and Its Effect on Esthetics. a Case Series Study
Brief Title: Implant Placement in Horizontally Deficient Maxillary Aesthetic Zone With Simultaneous Soft Tissue Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Maher Hakeem, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1975
Record Dates: First submitted 2022-02-02; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Implant or Graft; Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with missing teeth in maxillary aesthetic zone (Other)
  Interventions: Procedure: implant placement with simultaneous soft tissue augmentation

INTERVENTIONS:
Procedure: implant placement with simultaneous soft tissue augmentation — implant placement with simultaneous soft tissue augmentation using De-epithelialized free gingival graft and immediate temporization in the maxillary aesthetic zone .

SUMMARY:
Tooth extraction in maxillary esthetic zone is accomplished with great dimensional changes of the alveolar ridge, different procedures have been tested to compensate these dimensional alteration, such as Hard bone augmentation, Soft tissue augmentation Or augmentation of both together. Hence, the present study aimed to evaluate pink esthetic score, clinical implant stability and bucco-palatal dimensional changes in the maxillary esthetic zone treated by implant placement with simultaneous soft tissue augmentation using de-epithelialized free gingival graft.

ELIGIBILITY:
Inclusion Criteria:

* Patient of both sexes with missing teeth in the maxillary aesthetic zone.

Exclusion Criteria:

* Patients with systemic disease that may affect bone quality or bone healing.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
pink esthetic score | 6 month
  pink esthetic score evaluated pre-operative and 6 month post-operative (PES scale 0-1-2 , ''2'' the best , ''0'' the worst

SECONDARY OUTCOMES:
Implant stability quotient | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt